CLINICAL TRIAL: NCT00876993
Title: A Phase I Study Of Irinotecan and Bevacizumab With Temozolomide in Children With Recurrent/Refractory Central Nervous System Tumors
Brief Title: Study of Irinotecan and Bevacizumab With Temozolomide in Refractory/Relapsed Central Nervous System (CNS) Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Collaborators: The V Foundation (Other); Brain Tumor Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CNS-001
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Central Nervous System Tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Bevacizumab; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose Level 0 (Experimental): Bevacizmuab 10 mg/kg IV Irinotecan 125 mg/m^2 IV Temozolomide 75 mg/m^2 PO
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide
- Dose Level 1 (Experimental): Bevacizmuab 10 mg/kg IV Irinotecan 125 mg/m^2 IV Temozolomide 125 mg/m^2 PO
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide
- Dose Level 2 (Experimental): Bevacizmuab 10 mg/kg IV Irinotecan 125 mg/m^2 IV Temozolomide 175 mg/m^2 PO
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide
- Dose Level 3 (Experimental): Bevacizmuab 10 mg/kg IV Irinotecan 125 mg/m^2 IV Temozolomide 200 mg/m^2 PO
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide
- Dose Level 4 (Experimental): Bevacizmuab 10 mg/kg IV Irinotecan 150 mg/m^2 IV Temozolomide 200 mg/m^2 PO
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10 mg/kg IV on day 1 and day 15 of a 28 day cycle
  Other Names: Irinotecan and temozolomide
Drug: Irinotecan — Irinotecan 125 mg/m2 on day 1 and day 15 of a 28 day course given IV for the first 3 dose levels. If the Maximum Tolerated Dose of temozolomide is not reached at dose level 3, then dose level 4 will be an escalation of irinotecan to 150mg/m2.
  Other Names: Bevacizumab and temozolomide
Drug: Temozolomide — For the first cohort (dose level 0) of patients, dosing is 75 mg/m2/day day 1-5 of a 28 day course given PO for the first course. Doses will be escalated according to standard phase I dose escalation criteria. Dose levels are as follows (Dose level 1 = 125mg/m2, Dose level 2 = 175mg/m2, Dose levels 3 and 4 = 200 mg/m2)
  Other Names: Bevacizumab and irinotecan

SUMMARY:
Bevacizumab, irinotecan, and temozolomide are three agents shown to have promising activity in a variety of central nervous system tumors. No prospective studies have been published or are currently in progress within the major consortiums with this combination of drugs. Brain tumors are the second most common cause of cancer in pediatrics and the leading cause of cancer death in children. For children with High Grade Gliomas or with relapsed/refractory brain tumors, new agents in new combinations are needed. Historical data shows that newly diagnosed high grade gliomas 5 year progression free survival is 28-42%. Recurrent malignant gliomas median survival is 3-9 months. Recurrent medulloblastoma's 2 years survival is 9%. This study is a phase I study designed to provide an objective observation of toxicity and establish a maximum tolerated dose of this combination. In addition, this study will observe the response of children with relapsed or refractory central nervous system tumors.

DETAILED DESCRIPTION:
Bevacizumab dosing is 10 mg/kg on day 1 and day 15 of a 28 days course given IV.

Irinotecan dosing is 125 mg/m2 on day 1 and day 15 of a 28 day course given IV for the first 3 dose levels. If the MTD of temozolomide is not reached at dose level 3, then dose level 4 will be an escalation of irinotecan to 150 mg/m2.

For dose level 0 Temozolomide, dosing is 75 mg/m2/day day 1-5 of a 28 day course given PO. Doses will be escalated according to standard phase I dose escalation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Medulloblastomas, high-grade glioma, low-grade glioma, and ependymoma are eligible. Other central nervous system tumors may be considered for treatment at discretion of investigator. Pathology is required unless diffuse intrinsic pontine glioma or optic pathway tumor.
* The patient should have failed first line therapy and be considered refractory, relapsed, or recurrent. Exceptions are high grade gliomas including brain stem gliomas.
* Age 18 months though age 23 years are eligible for this protocol.
* The patient may have received any of the agents, but not in this combination. Patients will not be eligible if they have received the combination of bevacizumab and IV irinotecan as prior therapy. They will not be eligible if they had progressive disease on any of these agents. Investigator discretion may also be used.
* Bone marrow should be recovered from prior therapy with ANC >1500 and platelets >100,000.
* Serum creatinine should be less than institutional upper limit of norm.
* ALT/AST <3 times normal and bilirubin <1.5 times normal.
* Neurologic symptoms should be stable for 1 week with stable or decreasing doses of steroids.
* Patients should not be pregnant or breast feeding.

Exclusion Criteria:

* Patients with bleeding disorders or on anticoagulants.
* Uncontrolled hypertension.
* Other risks of bleeding determined on individual basis.
* Patients receiving enzyme inducing anticonvulsants.
* Patients with significant cardiac or pulmonary dysfunction that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results.
* For patients receiving bevacizumab, those who have had surgical procedures should not receive bevacizumab within 28 days of a major procedure, 14 days of an intermediate procedure and 7 days of a minor procedure. Lumbar punctures or placement of PICC lines are not considered minor procedures and may occur at any time prior to or during therapy.

Ages: 18 Months to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2008-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Stapleton, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will determine after further data analysis

REFERENCES:
- [Derived] Metts J, Harrington B, Salman E, Bradfield SM, Flanary J, Mosha M, Amankwah E, Stapleton S. A phase I study of irinotecan and temozolomide with bevacizumab in children with recurrent/refractory central nervous system tumors. Childs Nerv Syst. 2022 May;38(5):919-928. doi: 10.1007/s00381-022-05479-7. Epub 2022 Mar 8. PMID 35260913

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Dose Level 1; Cohort 3 - Dose Level 1; Cohort 5 - Dose Level 1: Bevacizmuab 10 mg/kg IV days 1 and 15 Irinotecan 125 mg/m^2 IV days 1 and 15 Temozolomide 125 mg/m^2 PO days 1-5 28 day cycle
- Cohort 2 - Dose Level 0: Bevacizmuab 10 mg/kg IV days 1 and 15 Irinotecan 125 mg/m^2 IV days 1 and 15 Temozolomide 75 mg/m^2 PO days 1-5 28 day cycle
- Cohort 4 - Dose Level 2: Bevacizmuab 10 mg/kg IV days 1 and 15 Irinotecan 125 mg/m^2 IV days 1 and 15 Temozolomide 175 mg/m^2 PO days 1-5 28 day cycle
Period: Overall Study
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1
Started (Began at Dose Level (DL) 1, next was DL 0 (de-escalation), followed by DL1, DL 2, finished at DL 1.) | 5 | 6 | 5 | 5 | 5
Completed | 4 | 6 | 3 | 5 | 3
Not Completed | 1 | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1 | Total
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 26
Age, Continuous [Mean (Full Range); unit: years] | 9.2 [5 to 14] | 8.5 [2 to 18] | 11.4 [4 to 22] | 9.8 [3 to 17] | 10.6 [6 to 14] | 9.8 [2 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 2 | 0 | 8
  Male | 3 | 5 | 2 | 3 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 2 | 1 | 3 | 4 | 3 | 13
  Unknown or Not Reported | 2 | 5 | 1 | 1 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 1 | 1 | 6
  White | 5 | 2 | 3 | 3 | 3 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 5 | 5 | 5 | 26
Diagnosis [Count of Participants; unit: Participants]
  Medulloblastoma | 0 | 0 | 1 | 0 | 1 | 2
  High Grade Glioma | 3 | 2 | 2 | 2 | 2 | 11
  Low Grade Glioma | 1 | 1 | 1 | 2 | 1 | 6
  Choroid Plexus Tumors | 1 | 0 | 0 | 0 | 0 | 1
  Ependymoma | 0 | 2 | 0 | 0 | 0 | 2
  PNET | 0 | 1 | 0 | 1 | 1 | 3
  Other | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Number of Adverse Events
Description: Collect and grade the all of the adverse events to evaluate for safety. This data was collected for the first 2 cycles for each participant.
Time Frame: Two 28-day cycles
Measure: Number; unit: Adverse events
Groups:
- Cohort 4 - Dose Level 2: BBevacizmuab 10 mg/kg IV days 1 and 15 Irinotecan 125 mg/m^2 IV days 1 and 15 Temozolomide 175 mg/m^2 PO days 1-5 28 day cycle
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1
Number analyzed (Participants) | 4 | 6 | 3 | 5 | 3
Adverse events
  Grade 1 adverse events | 4 | 6 | 3 | 5 | 3
  Grade 2 adverse events | 4 | 3 | 3 | 5 | 2
  Grade 3 adverse events | 3 | 1 | 1 | 4 | 1
  Grade 4 adverse events | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Best Response of Children With Recurrent or Refractory Central Nervous System Tumors With This Combination of Chemotherapy Agents.
Description: Best response by MRIs per definitions in the protocol (complete response, partial response, stable disease, progressive disease). MRI's were obtained every 2 cycles and the best response was reported.
Time Frame: Every 2 cycles up to 24 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1
Number analyzed (Participants) | 4 | 6 | 3 | 5 | 3
Participants
  Complete Response | 0 | 0 | 0 | 1 | 0
  Partial Response | 1 | 1 | 1 | 3 | 0
  Stable Disease | 3 | 3 | 0 | 1 | 3
  Progressive Disease | 0 | 2 | 2 | 0 | 0

3. Secondary Outcome: 2 Year Event Free Survival With Children Treated With This Regimen.
Description: 2 year actual event free survival.with children treated with this protocol
Time Frame: 2 year
Measure: Number; unit: Count of participants
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1
Number analyzed (Participants) | 4 | 6 | 3 | 5 | 3
Count of participants | 4 | 6 | 3 | 5 | 3

4. Secondary Outcome: To Provide Safety and Efficacy Data for to Recommend Further Larger Studies.
Description: Number participants with grade 3 and 4 hematologic and non-hematologic toxicities. All toxicities are for end of cycle 2.
Time Frame: Two 28 day cycles
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5 - Dose Level 1: BBevacizmuab 10 mg/kg IV days 1 and 15 Irinotecan 125 mg/m^2 IV days 1 and 15 Temozolomide 125 mg/m^2 PO days 1-5 28 day cycle
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1
Number analyzed (Participants) | 4 | 6 | 3 | 5 | 3
Participants
  Grade 3 & 4 Blood/Bone Marrow | 2 | 0 | 0 | 1 | 1
  Grade 3 & 4 Gastrointestinal | 0 | 0 | 1 | 1 | 0
  Grade 3 & 4 Metabolic/Laboratory | 0 | 0 | 0 | 1 | 0
  Grade 3 & 4 Musculoskelatal/Soft Tissue | 0 | 0 | 0 | 1 | 0
  Grade 3 & 4 Neurology | 1 | 0 | 0 | 3 | 0
  Grade 3 & 4 Pain | 1 | 0 | 0 | 2 | 0
  Grade 3 & 4 Vascular | 0 | 1 | 0 | 0 | 0
  Grade 3 & 4 Other | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Two 28 day cycles for each participant
Arm/Group | Cohort 1 - Dose Level 1 | Cohort 2 - Dose Level 0 | Cohort 3 - Dose Level 1 | Cohort 4 - Dose Level 2 | Cohort 5 - Dose Level 1
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/6 | 1/5 | 4/5 | 1/5
Other Adverse Events (participants affected / at risk) | 4/5 | 1/6 | 2/5 | 3/5 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Dose Level 1 (N=5) | Cohort 2 - Dose Level 0 (N=6) | Cohort 3 - Dose Level 1 (N=5) | Cohort 4 - Dose Level 2 (N=5) | Cohort 5 - Dose Level 1 (N=5)
Neurology, other - pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombus - embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GI illness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurologic deficits (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shunt malfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dystonic reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hemolytic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Dose Level 1 (N=5) | Cohort 2 - Dose Level 0 (N=6) | Cohort 3 - Dose Level 1 (N=5) | Cohort 4 - Dose Level 2 (N=5) | Cohort 5 - Dose Level 1 (N=5)
Leukocytes (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 3 and 4
Neutrophils (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Grade 3 and 4
Lymphocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ALT/AST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombus (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope/Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No